CLINICAL TRIAL: NCT03502304
Title: Concurrent Training and Prediabetes Comorbidities: An Analysis of Non-responders Using Clinical Cutoff Points
Brief Title: Concurrent Training and Prediabetes Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Universidad de Los Lagos (Other); Healthcare Center Tomas Rojas (Other); Universidad del Rosario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9042018
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Disturbance
Keywords: Metabolic syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Endurance Training

STUDY DESIGN:
Intervention Model Description: Behavioral
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): No-exercise
  Interventions: Behavioral: Endurance training plus resistant training
- Endurance training plus resistant training (Experimental): To concurrent training (endurance training plus resistant training, RT) program will be use cycle ergometers adapted for obese adults (OXFORDTM, model BE2601, OXOFORD Inc, Santiago, Chile) were used. Prior to the CT intervention, all subjects were familiarized (during 3 sessions) with the training protocols. The CT intervention included 3 weekly sessions of both ET and RT. The core part of each session included RT followed by ET exercises (for 50 and 30 minutes, respectively) and was preceded and followed by a 5-minute warm-up and cool-down with callisthenic movements.
  Interventions: Behavioral: Endurance training plus resistant training

INTERVENTIONS:
Behavioral: Endurance training plus resistant training — CT in women with prediabetes and co-morbidities associated. Exercise will be performed at three sessions per week. Post statistical analyses will be including analyses by the 2 groups proposed. All sessions will be supervised by an exercise physiologist during 20-weeks.

SUMMARY:
Despite exercise training decrease blood fasting glicaemy in 'average' terms, there is a wide inter-individual variability after exercise training explored mainly in adults but not in adults with prediabetes comorbidities. Thus, is yet unknown the effects and influence of the concurrent training (CT) eliciting responders (R) and non-responders (NR) cases (i.e., percentage of subjects who experienced a non-change/worsened response after training in some metabolic outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Interested in improving health and fitness.

Exclusion Criteria:

* Cardiovascular contraindications to exercise,
* History of stroke, asthma or chronic obstructive pulmonary disease,
* Muscle-skeletal disorders, and
* Smoking.
* A compliance rate to the exercise program ≥ 70% was required for the participants in the intervention group to be included in the statistical analyses.

Ages: 30 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in fasting glucose
Lipoproteins | Baseline and 20-weeks immediately after the interventions ends
  Change from baseline in lipoproteins

SECONDARY OUTCOMES:
Body mass | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in body mass
Waist circumference | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in waist circumference
Fat mass | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in fat mass
Lean mass | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in lean mass
Heart rate at rest | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in heart rate at rest
Six minutes walking test | Baseline and 20-weeks immediately after the interventions ends
  Change from Baseline in six minutes walking test

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Alvarez, PhD, Principal Investigator — Universidad de Los Lagos
Locations (1):
- Cristian Alvarez, Los Lagos, Osorno, Chile

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03502304/Prot_SAP_000.pdf